CLINICAL TRIAL: NCT03700476
Title: Sintilimab (PD-1 Antibody) and Chemoradiotherapy in Locoregionally-advanced Nasopharyngeal Carcinoma: a Randomized, Multicenter, Phase 3 Trial
Brief Title: Sintilimab (PD-1 Antibody) and Chemoradiotherapy in Locoregionally-advanced Nasopharyngeal Carcinoma
Acronym: CONTINUUM
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-FXY-135-FLK
Record Dates: First submitted 2018-10-03; First posted 2018-10-09 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms | interventions — sintilimab; spartalizumab; Gemcitabine; Cisplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sintilimab arm (Experimental): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT. Sintilimab 200mg will be given every 3 weeks for 12 cycles, started on day 1 of induction chemotherapy.
  Interventions: Drug: Sintilimab; Drug: Gemcitabine; Drug: Cisplatin; Radiation: intensity-modulated radiotherapy
- Chemoradiation arm (Active Comparator): Patients will receive induction chemotherapy with gemcitabine (1g/m2, d1 & 8 of every cycle) and cisplatin (80mg/m2, d1 of every cycle), every 3 weeks for 3 cycles before radiation. Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy in 33 fractions will be given. Concurrent cisplatin of 100mg/m2 will be administered every 3 weeks for 2 cycles during IMRT.
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Radiation: intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Sintilimab — Sintilimab 200mg will be given every 3 weeks for 12 cycles, started on day 1 of induction chemotherapy.
  Other Names: IBI308; PD-1 antibody
  Arms: Sintilimab arm
Drug: Gemcitabine — Gemcitabine 1g/m2, d1 & 8 of every cycle, every 3 weeks for 3 cycles before radiation.
Drug: Cisplatin — Induction cisplatin 80mg/m2, every 3 weeks for 3 cycles before radiation; Concurrent cisplatin 100mg/m2, every 3 weeks for 2 cycles during radiation
  Other Names: DDP
Radiation: intensity-modulated radiotherapy — Definitive intensity-modulated radiotherapy (IMRT) of 6996cGy will be given in 33 fractions.
  Other Names: IMRT

SUMMARY:
The CONTINUUM trial plans to enroll patients with stage III-IVA (AJCC 8th, except T3N0-1 or T4N0) locoregionally-advanced nasopharyngeal carcinoma (LANPC). Patients will be randomized in a 1:1 ratio to receive 3 cycles of induction chemotherapy with gemcitabine and cisplatin and concurrent cisplatin-radiation or the same regimen plus Sintilimab. All patients will receive intensity-modulated radiotherapy (IMRT). Sintilimab will begin on day 1 of induction chemotherapy and continue every 3 weeks for 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically confirmed nasopharyngeal carcinoma.
2. Tumor staged as III-IVA (AJCC 8th, except T3N0-1 or T4N0).
3. Eastern Cooperative Oncology Group performance status ≤1.
4. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.
5. Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN.
6. Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).
7. Patients must be informed of the investigational nature of this study and give written informed consent.
8. Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug.

Exclusion Criteria:

1. Age > 65 or < 18.
2. Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA >1×10e3 copies/ml or 200IU/ml
3. Hepatitis C virus (HCV) antibody positive
4. Has active autoimmune disease, except type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia).
5. Has any condition that required systemic corticosteroid (equivalent to prednisone >10mg/d) or other immunosuppressive therapy within 28 days before informed consent. Patients received systemic corticosteroid equivalent to prednisone ≤10mg/d, inhale or topical corticosteroid will be allowed.
6. Has a known history of active TB (bacillus tuberculosis) within 1 year; patients with adequately treated active TB over 1 year ago will be allowed.
7. Has a known history of interstitial lung disease.
8. Has received a live vaccine within 30 days before informed consent or will receive a live vaccine in the near future.
9. Is pregnant or breastfeeding.
10. Prior malignancy within 5 years, except in situ cancer, adequately treated non-melanoma skin cancer, and papillary thyroid carcinoma.
11. Has known allergy to large molecule protein products or any compound of sintilimab.
12. Has a known history of human immunodeficiency virus (HIV) infection.
13. Any other condition, including symptomatic heart failure, unstable angina, myocardial infarction, active infection requiring systemic therapy, mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 425 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | 3 years
  calculated from randomization to the date of locoregional recurrence, distant metastasis, or death from any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival (OS) | 3 years
  calculated from randomization to the date of death from any cause.
Distant metastasis-free survival (DMFS) | 3 years
  calculated from randomization to the date of first distant metastasis, or death from any cause, whichever occurred first.
Locoregional recurrence-free survival (LRFS) | 3 years
  calculated from randomization to the date of locoregional persistence, 1st locoregional recurrence, or death from any cause, whichever occurred first.
Adverse events (AEs) and serious adverse events (SAEs) | 3 years
  Graded according to CTCAE V5.0.
Quality of life (QoL) | 3 years
  The change of QoL from randomization to the start of radiotherapy, the end of radiotherapy, 34 weeks (at the end of sintilimab treatment in the sintilimab arm and the corresponding timepoint in the chemoradiation arm), 2 years and 3 years after randomization. The EORTC QoL questionnaire-C30 (EORTC QLQ-C30）version 3.0 will be used. This questionnaire comprises 30 questions, 24 of which are aggregated into nine multi-question scales, that is, five functioning scales (e.g., physical), three symptom scales (e.g., fatigue) and one global health status scale. The remaining six single-question (e.g., dyspnoea) scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual.
Event-free survival (EFS) within different subgroups | 3 years
  analyses for EFS will be performed within the following subgroups: Epstein-Barr virus (EBV) DNA (<4000copies/ml vs. ≥4000copies/ml), different PD-L1 expression levels (<1% vs. ≥1%), tertiary lymphoid structure (+ vs. -), age, gender, performance status, T category, N category, and stage (III vs. IVA).

OTHER OUTCOMES:
The association of circulation autoimmune antibodies with immune-related adverse events | 1 year
The association of circulation cytokines, chemokines, and growth factors/regulators with immune-related adverse events | 1 year
The association of gene expression with the efficacy of sintilimab | 3 years
  RNA sequencing will be conducted using baseline tumor samples.
The association of cell populations with the efficacy of sintilimab | 3 years
  Multiplex Immunofluorescence will be conducted to assess tumor and immune-related markers in baseline tumor samples.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, MD, Principal Investigator — Sun Yat-sen University
Locations (9):
- China (9):
  - First People's Hospital of Foshan, Foshan, Guangdong
  - Panyu central hospital, Guangzhou, Guangdong
  - SUN YAT-SEN UNIVERSITY cANCER CENTER, Guangzhou, Guangdong
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Xijing Hospital, Fourth Military Medical University, Xi’an, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
Complete de-identified patient data set
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: For 2 years started from 12 months after publication of the primary trial report.
Access Criteria: Authoritative researchers who provide a methodologically sound proposal for individual participant data meta-analysis.

REFERENCES:
- [Derived] Zou SQ, Huang CL, Zhang JJ, Li Z, Xiao XT, Cheng YZ, Shen JY, Wu DH, Lv JW, Tang LL, Sun Y, Li JB, Liu X, Ma J, Li WF, Chen YP. Association of anti-PD-1 therapy with severe radiation-induced oral mucositis: A retrospective cohort study and validation in the CONTINUUM trial. Med. 2025 Oct 10;6(10):100770. doi: 10.1016/j.medj.2025.100770. Epub 2025 Jul 11. PMID 40651471
- [Derived] Huang SW, Jiang W, Xu S, Zhang Y, Du J, Wang YQ, Yang KY, Zhang N, Liu F, Zou GR, Jin F, Wu HJ, Zhou YY, Zhu XD, Chen NY, Xu C, Qiao H, Liu N, Sun Y, Ma J, Liang YL, Liu X. Systemic longitudinal immune profiling identifies proliferating Treg cells as predictors of immunotherapy benefit: biomarker analysis from the phase 3 CONTINUUM and DIPPER trials. Signal Transduct Target Ther. 2024 Oct 23;9(1):285. doi: 10.1038/s41392-024-01988-w. PMID 39438442
- [Derived] Liu X, Zhang Y, Yang KY, Zhang N, Jin F, Zou GR, Zhu XD, Xie FY, Liang XY, Li WF, He ZY, Chen NY, Hu WH, Wu HJ, Shi M, Zhou GQ, Mao YP, Guo R, Sun R, Huang J, Liang SQ, Wu WL, Su Z, Li L, Ai P, He YX, Zang J, Chen L, Lin L, Huang SH, Xu C, Lv JW, Li YQ, Hong SB, Jie YS, Li H, Huang SW, Liang YL, Wang YQ, Peng YL, Zhu JH, Zang SB, Liu SR, Lin QG, Li HJ, Tian L, Liu LZ, Zhao HY, Lin AH, Li JB, Liu N, Tang LL, Chen YP, Sun Y, Ma J. Induction-concurrent chemoradiotherapy with or without sintilimab in patients with locoregionally advanced nasopharyngeal carcinoma in China (CONTINUUM): a multicentre, open-label, parallel-group, randomised, controlled, phase 3 trial. Lancet. 2024 Jun 22;403(10445):2720-2731. doi: 10.1016/S0140-6736(24)00594-4. Epub 2024 May 30. PMID 38824941